CLINICAL TRIAL: NCT02277730
Title: A Novel Closed-loop Integrated System for the Maintenance of Haemodynamic Stability to Improve Perioperative Outcome During Spinal Anaesthesia for Caesarean Section
Brief Title: A Novel Closed-loop Integrated System for the Maintenance of Haemodynamic Stability
Acronym: DIVA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHF/CTG047/2012
Record Dates: First submitted 2014-10-26; First posted 2014-10-29 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2017-08

CONDITIONS: Hypotension
Keywords: Hypotension
MeSH Terms: conditions — Hypotension | interventions — Phenylephrine; Vasoconstrictor Agents; Ephedrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- vasopressor delivery automated system (Experimental): vasopressor delivery automated system administering phenylephrine and ephedrine using a 2 step algorithm vasopressor delivery technique
  Interventions: Device: vasopressor delivery automated system; Drug: phenylephrine; Drug: ephedrine
- manual vasopressor delivery (Active Comparator): manual bolus delivering phenylephrine and ephedrine using a 2 step algorithm vasopressor delivery technique
  Interventions: Drug: phenylephrine; Drug: ephedrine; Device: manual vasopressor delivery

INTERVENTIONS:
Device: vasopressor delivery automated system — vasopressor delivery using phenylephrine and ephedrine
  Other Names: vasopressor delivery technique
  Arms: vasopressor delivery automated system
Drug: phenylephrine
  Other Names: vasopressor
Drug: ephedrine
  Other Names: vasopressor
Device: manual vasopressor delivery
  Arms: manual vasopressor delivery

SUMMARY:
Hypotension occurs commonly during spinal anaesthesia for caesarean section with maternal and fetal adverse effects. The investigators developed a double-vasopressor automated system incorporating continuous non-invasive haemodynamic monitoring using NexfinTM with a two-step algorithm.

DETAILED DESCRIPTION:
Hypotension occurs commonly during spinal anaesthesia for caesarean section with maternal and fetal adverse effects. We developed a double-vasopressor automated system incorporating continuous non-invasive haemodynamic monitoring using Nexfin cardiac output monitor with a two-step algorithm. The system delivered phenylephrine 25 mcg or ephedrine 2 mg (if heart rate<60 beats.min-1) every 30 seconds when systolic blood pressure was between 90-100% of baseline. The system delivered phenylephrine 50 mcg or ephedrine 4 mg (if heart rate<60 beats.min-1) every 30 seconds when systolic blood pressure was <90% of baseline.

A randomised controlled trial will be done to compare with manual bolus technique. With the manual bolus technique, phenylephrine 50mcg or ephedrine 4mg (if heart rate<60 beats.min-1) every 60 seconds when systolic blood pressure was between 90-100% of baseline. The system delivered phenylephrine 100mcg or ephedrine 8mg (if heart rate<60 beats.min-1) every 60 seconds when systolic blood pressure was <90% of baseline.

ELIGIBILITY:
Inclusion Criteria:

* age 21-45 years old,
* weight 40-90 kg,
* height 145-170 cm

Exclusion Criteria:

* contraindications to spinal anaesthesia,
* allergy to drugs used in the study, and
* those with uncontrolled medical conditions such as hypertension, diabetes mellitus, and cardiovascular disease

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 252 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Hypotension | 1 day
  Systolic blood pressure less than 80% of baseline systolic blood pressure

SECONDARY OUTCOMES:
Hypertension | 1 day
  Systolic blood pressure more than 120% of baseline systolic blood pressure
Nausea and vomiting | 1 day
  Nausea and vomiting during Caesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Ban L Sng, FANZCA, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Du EW, Tan HS, Tan CW, Sultana R, Sng BL. Heart rate variability and haemodynamic factors associated with hypotension during spinal anaesthesia for caesarean delivery: A case-control study. Eur J Anaesthesiol. 2022 Mar 1;39(3):219-226. doi: 10.1097/EJA.0000000000001551. PMID 34101716
- [Derived] Sng BL, Du W, Lee MX, Ithnin F, Mathur D, Leong WL, Sultana R, Han NR, Sia ATH. Comparison of double intravenous vasopressor automated system using nexfin versus manual vasopressor bolus administration for maintenance of haemodynamic stability during spinal anaesthesia for caesarean delivery: A randomised double-blind controlled trial. Eur J Anaesthesiol. 2018 May;35(5):390-397. doi: 10.1097/EJA.0000000000000779. PMID 29373334